CLINICAL TRIAL: NCT06612866
Title: Determination of the Biological Activity of Enriched Serums on Healthy Volunteers After Consumption of the Kera-Diet® Ingredient, CnC2024 - Kera-Diet®
Brief Title: Determination of the Biological Activity of Enriched Serums on Healthy Volunteers After Consumption of the Kera-Diet® Ingredient
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BCF Life Sciences (Industry)
Collaborators: Clinic'n'Cell (Other); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-A01011-46
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Kera-Diet treatment (Other)
  Interventions: Dietary Supplement: Keratin hydrolysate

INTERVENTIONS:
Dietary Supplement: Keratin hydrolysate — The clinical study will be conducted in two phases. The first phase will aim at characterizing the metabolites present in human serum after consumption of the Kera-Diet® ingredient and at determining the overall absorption peak of the tested ingredient. The second phase will involve collecting sera enriched with metabolites at the absorption peak, following the ingestion of the ingredient. Subsequently, the final objective will be to characterize the influence of these sera enriched with metabolites of interest on the behavior of human skin cell and intestinal epithelial cell cultures.

SUMMARY:
The main objective of this study is, after collecting serum enriched with metabolites of interest resulting from the ingestion of the Kera-Diet® food supplement, to determine the influence of these sera enriched with circulating metabolites (versus naïve sera) on the behavior of human cell cultures, placed under stress conditions or not, in order to evaluate the benefit of these metabolites in maintaining cellular functions.

ELIGIBILITY:
Main inclusion Criteria:

* Liver function tests within reference norms.
* Kidney function tests within reference norms.
* Complete blood count (CBC) within reference norms.
* C-reactive protein (CRP) within reference norms.
* Blood pressure compatible with study requirements.
* Non-smoker or occasional smoker (max 5 cigarettes/day or max 10 ml per week of e-liquid with a nicotine concentration of 3 mg/ml).
* Max 5 hours of intense sports per week.
* Weight ≥ 60 kg.
* BMI between 20 and 28 kg/m² (exclusive).

Main exclusion Criteria:

* Any type of vaccination within the past month.
* Alcohol consumption exceeding WHO standards (Sup. 3 drinks per day for men).
* Ongoing treatment (medication, dietary supplement, or probiotic) and within the four weeks prior to inclusion.
* Known pathology (including seasonal).
* Allergy to the study product, particularly to keratin or certain amino acids.
* Individuals following a diet unsuitable for the study (e.g., vegetarian, vegan, or plant-based diets).
* Change in eating habits within the 4 weeks prior to inclusion.
* Medical and/or surgical history deemed incompatible with the trial by the investigator or their representative.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Determination of the influence of human serums enriched with circulating metabolites on human cell cultures | Determination of the absorption peak: kinetics will be determined by a blood draw at different time points (T0, T5, T10, T20, T30, T45, T60, T80, T100, T120, T140, T180, T240 minutes) over the 4 hours following the ingestion of the study product
  Determination of the influence of human serums enriched with circulating metabolites (versus naïve serums) on the behavior of human cell cultures exposed or not to stress conditions in order to evaluate the benefit of these metabolites in maintaining cellular functions.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- University Hospital, Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No